CLINICAL TRIAL: NCT04784572
Title: Assessment of Pain During Intramuscular Injection Delay in Adult Psychiatry
Acronym: evadoulim
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Principal Investigator, Dominique JANUEL, HEAD OF THE UNIT OF CLINICAL RESEARCH, Centre hospitalier de Ville-Evrard, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10477M-EVADOULIM
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Delayed Antipsychotic Treatment, Pharmacological Factors and Individual Factors
Keywords: pain -injection

STUDY DESIGN:
Intervention Model Description: The group will have a first injection delay and then a second injection delay.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- First injection delay and second injection delay (Other): During the first injection, the patient will make 3 scales: END, EVAF and insight and there will be an assessment of induration, redness and swelling done with nurses.
  During the second injection, the patient will perform the END and EVAF scale and then follow up with a maintenance
  Interventions: Other: first injection delay and second injection delay

INTERVENTIONS:
Other: first injection delay and second injection delay — During the first injection, the patient will make END scale for 5 seconds, EVAF scale for 10 seconds and insight scale for 5 minutes.
  The second injection the patient will make END scale for 5 seconds and EVAF scale for 10 seconds and then a maintenance.

SUMMARY:
Since psychiatry is still too often confronted with a dichotomy between psyche and soma, the assessment of pain and anxiety at RMI is still rarely done (Willer et al., 1982). The objective of this exploratory study is to evaluate the influence of pharmacological factors (type of injected molecules, injection frequency, injection site, treatment duration, treatment dose, time since last injection) and individual about the pain perceived when injecting antipsychotic therapy (diagnosis, sex, age, weight, duration of illness, level of anxiety, psychiatric and somatic comorbidity, insight). In the future, this study will develop a suitable procedure to limit pain and anxiety during RMI. Taking these dimensions into account will probably allow a better compliance of patients for this type of care, and thus a decrease in the number of relapses in the long term.

ELIGIBILITY:
Inclusion Criteria:

* Patients (Males, Females)
* Over the age of 18
* Hospitalized or outpatient
* Patient affiliated with social security, State Medical Aid (AME)
* With prescription of antipsychotic delay by intramuscular injection
* French language mastered
* Given oral consent to pass the self-assessment scales

Exclusion Criteria:

* Patients on long-term analgesic treatment, daily
* Patients with chronic pain with or without analgesic treatment
* Patient not communicating
* Pregnant woman, parturint and nursing mother
* Person deprived of liberty by judicial or administrative decision
* Minor and person subject to legal protection: guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The Digital Scale of Pain (END) | At the first visit during the first injection of treatment delay . It will take 5 seconds
  This scale will assess pain at the injection site before and after intramuscular injection of neuroleptic treatment delay.
  This scale ranges from 0 (none pain) to 10 (worst possible pain). It will only take 5 seconds for the subject. This scale has good concurrent validity because it is highly correlated with others pain measurement tools (Haefeli & Elfering, 2006), including the analog visual scale of pain (r=0.95; p<0.001; Bahreini et al., 2015).
The Digital Scale of Pain (END) | At the second visit during the first injection of treatment delay . It will take 5 seconds
  This scale will assess pain at the injection site before and after intramuscular injection of neuroleptic treatment delay.
  This scale ranges from 0 (none pain) to 10 (worst possible pain). It will only take 5 seconds for the subject. This scale has good concurrent validity because it is highly correlated with others pain measurement tools (Haefeli & Elfering, 2006), including the analog visual scale of pain (r=0.95; p<0.001; Bahreini et al., 2015).
Facial Anxiety Visual Scale (EVAf) | At the first visit during the first injection of treatment delay . It will take10 seconds.
  This scale Assess patient anxiety before and after intramuscular injection of delayed neuroleptic therapy. It was developed by Cao et al., (2017).
  It is a self-assessment scale of the severity of anxiety representing facial expression during anxiety.
  Six faces represent different expressions of anxiety: "No anxiety", "Mild anxiety", Mild to Moderate Anxiety, Moderate Anxiety, Moderate to High Anxiety, and High Anxiety.
Facial Anxiety Visual Scale (EVAf) | At the second visit during the first injection of treatment delay . It will take 10 seconds.
  This scale Assess patient anxiety before and after intramuscular injection of delayed neuroleptic therapy. It was developed by Cao et al., (2017).
  It is a self-assessment scale of the severity of anxiety representing facial expression during anxiety.
  Six faces represent different expressions of anxiety: "No anxiety", "Mild anxiety", Mild to Moderate Anxiety, Moderate Anxiety, Moderate to High Anxiety, and High Anxiety.
Insight scale (BIS) | At the first visit during the first injection of treatment delay . It will take5 minutes.
  This scale will assess the knowledge of the disease, the insight of patients, prior to intramuscular injection of neuroleptic therapy delay to Visit 1 (V1). This questionnaire developed by Birchwood et al. (1994), translated and validated in French by Linder and Favrod, (2006),will allow a quick self-assessment of the patient's insight. It consists of 8 items with a duration of 5 minutes. The person can choose between 3 answers for each item: "Agree", "In disagreement", "Uncertaine".
  The score is obtained by adding the score of the items:
  * Maximum score = 12 - Very good insight
  * 9 and above = good insight
  * Minimum score = 0 - No insight

CONTACTS AND LOCATIONS:
Locations (1):
- Ch Ville Evrard, Neuilly-sur-Marne, France

IPD SHARING:
Plan to Share IPD: Undecided